CLINICAL TRIAL: NCT04997044
Title: A Randomized Controlled Study Investigating the Effect of Designed Physical Training After Selective Dorsal Rhizotomy on Motor Function of Ambulant Children With Spastic Diplegia
Brief Title: Effect of Designed Physical Training After Selective Dorsal Rhizotomy on Motor Function of Ambulant Children With Spastic Diplegia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira Mahmoud Abd-elmonem, Amira Abd-elmonem, assist Prof. Physiacl therapy for pediatric department, faculty of physical therapy , Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: selective dorsal rhizotomy
Record Dates: First submitted 2021-08-04; First posted 2021-08-09 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Cerebral Palsy
Keywords: standard orthotic management; Selective dorsal rhizotomy; Bilateral Cerebral Palsy; Functional balance; Energy Cost of Walking; Functional capacity; Selective voluntary motor control:
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Other): control group
  Interventions: Other: Concomitant physical rehabilitation; Other: Standard Orthotic Management
- Experimental group (Experimental): selective dorsal rhizotomy group
  Interventions: Other: Concomitant physical rehabilitation; Other: Standard Orthotic Management; Other: selective dorsal rhizotomy

INTERVENTIONS:
Other: Concomitant physical rehabilitation — Children of this group will receive a regular exercise rehabilitation program including starching exercises, functional strength training and static and dynamic balance exercises.The program will be conducted by six licensed pediatric physical therapists for one hour/session, 3 times/week, and six successive months.
Other: Standard Orthotic Management — A custom-made articulating ankle foot orthosis was prescribed with a hinge at the level of the medial malleolus extends distally to the tip of the toes and proximally on the posterior surface of the leg to about 5 cm below the knee and secured straps. It is fabricated to permit free ankle dorsiflexion and lock the plantar flexion at 0 dorsiflexion. The splinting schedule started gradually for 2 h/day in the first month, 4 h/day in the second month to the entire wake-up time of the day.
Other: selective dorsal rhizotomy — The surgical procedures were tailored to each child according to preoperative assessment plan. All SDRs were performed by a single neurosurgeon through an osteoplastic laminotomy from L2 to L5 that left the facet joints intact.
  Arms: Experimental group

SUMMARY:
The management of cerebral palsy is complex and requires a multidisciplinary approach. Selective dorsal rhizotomy is a neurosurgical technique that aims to reduce spasticity in the lower limbs and improve motor function.

DETAILED DESCRIPTION:
the current study is designed to assess the effectiveness of Selective dorsal rhizotomy on motor function in ambulant children with spastic diplegia. therefore, A convenient sample of ambulant children with spastic diplegia will be allocated to two groups of equal numbers (control and experimental)

ELIGIBILITY:
Inclusion Criteria:

* CP, spastic diplegia
* 4-8 years of age
* The ability to walk with or without assistive devices typically on Level II-III on Gross Motor Function Classification System
* At least six months after the last Botulinum toxin A injection in the lower extremities
* Average intelligent quotient according to medical records for active participation
* Good trunk control with good antigravity strength of lower extremity on clinical examination.

Exclusionary criteria

* Ankle clonus; exaggerated deep tendon reflex in the legs
* Babinski sign
* Structural non-reducible deformities or musculoskeletal surgery in the lower extremities in the past 12 months
* Moderate to severe signs of dystonia, athetosis or ataxia.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Functional Balance | after 6 months and after 1 year (follow-up)
  The pediatric balance scale was used to assess the child's functional performance with total score is 56 and higher score representing a better performance.
Gross motor function | after 6 months and after 1 year (follow-up)
  The gross motor function measure-88 is used to evaluate the motor function with total score is 100 and higher scores representing a better performance.

SECONDARY OUTCOMES:
Selective voluntary motor control | after 6 months and after 1 year (follow-up)
  Selective motor control of lower extremity scale is used for assessment of motor control of the lower limb joints in children with spastic cerebral palsy with a maximum score of 20 points, 10 points for each limb.
Energy cost of walking | after 6 months and after 1 year (follow-up)
  The energy expenditure index (beats/meter) can be calculated as; walking heart rate (beats/min) minus resting heart rate (beats/ min) on walking velocity (meters/min).
Functional capacity | after 6 months and after 1 year (follow-up)
  The six-minute walking test is used to assess walking capacity in children with and without disabilities.

CONTACTS AND LOCATIONS:
Overall Officials: Hazem A Aly, Phd, Study Chair — PhD of physical therapy for pediatrics, faculty of physical therapyCairo university; Ahmed Rabie, Phd, Study Director — Department of neurosurgery, faculty of medicine , Alexandria university; Sara S Saad-Eldien, PhD, Principal Investigator — Cairo university, faculty of physical therapy
Locations (1):
- Amira Mahmoud Abd-elmonem, Giza, Egypt